CLINICAL TRIAL: NCT07388316
Title: Investigation of the Relationship Between Functional Improvement and Changes in Fine Manual Dexterity in Isolated Thumb Tendon Injuries
Brief Title: Functional Improvement and Fine Dexterity in Thumb Tendon Injuries
Status: Not yet recruiting | Type: Observational
Sponsor: Pamukkale University (Other)
Responsible Party: Principal Investigator, UMUT ERASLAN, Assistant Professor, Pamukkale University
Other Study IDs: E-60116787-020-808746
Record Dates: First submitted 2026-01-28; First posted 2026-02-05 (Actual); Last update posted 2026-02-06 (Actual); Status verified 2026-02

CONDITIONS: Thumb Injury; Tendon Injuries
Keywords: functional status; fine dexterity; thumb; tendon injury
MeSH Terms: conditions — Tendon Injuries | interventions — Surveys and Questionnaires; Restraint, Physical

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 24 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients diagnosed with isolated thumb tendon injuries at the hand level, who underwent surgical tre
  Interventions: Other: Questionnaire and Physical Exam

INTERVENTIONS:
Other: Questionnaire and Physical Exam — Joint range of motion, fine manual dexterity, reaction time, and grip strength will be assessed, and the Michigan Hand Outcomes Questionnaire will be administered to the patients.

SUMMARY:
Considering the thumb's contribution to fine dexterity and precision grip, this study aims to evaluate fine manual dexterity alongside functional outcomes following isolated thumb tendon injuries, and to examine the relationship between postoperative functional improvement and changes in fine manual dexterity.

ELIGIBILITY:
Inclusion Criteria:

* No history of neurological, orthopaedic, rheumatological, metabolic disease or surgery in the relevant extremity

Exclusion Criteria:

* Comorbid musculoskeletal-neurovascular injuries

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with surgically repaired isolated thumb tendon injuries
Sampling Method: Non-Probability Sample
Enrollment: 52 (Estimated)
Dates: Start 2026-02-26 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-03-01 (Estimated)

PRIMARY OUTCOMES:
Goniometric measurement | At postoperative 12th and 24th week
  Joint mobility will be measured in degrees (°) using a universal goniometer. Active flexion and extension of the Metacarpophalangeal (MCP) and Interphalangeal (IP) joints will be recorded. Higher degrees indicate better joint mobility.
Gross and fine grip strength | At postoperative 12th and 24th week
  Gross grip strength will be measured in kilograms (kg) using a Jamar Hand Dynamometer. Fine grip strength will be measured in kilograms (kg) using a Jamar Pinch gauge. Key pinch, tip-to-tip pinch, tripod pinch and pulp-to-pulp pinch strengths will be assessed. Patients will perform three maximum effort trials, and the mean value will be recorded. Higher values indicate greater strength.
Michigan Hand Outcomes Questionnaire | At postoperative 12th and 24th week
  he questionnaire covers 6 domains: overall hand function, activities of daily living, pain, work performance, appearance, and satisfaction. Total scores range from 0 to 100. For the pain domain, higher scores indicate more pain; for all other domains, higher scores indicate better hand function.
The O'Connor Finger Dexterity Test | At postoperative 12th and 24th week
  The unit of measure is the time in seconds required to complete the placement of pins in the board. Lower time values indicate better fine motor skill and manual dexterity.
The Nelson Hand Reaction Test | At postoperative 12th and 24th week
  The participant's reaction is measured by the distance the ruler falls before being caught measured in centimeters.Lower values (shorter distance) indicate faster reaction speed and better neuromuscular coordination.

CONTACTS AND LOCATIONS:
Locations (1):
- Pamukkale University, Denizli, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Starr HM, Snoddy M, Hammond KE, Seiler JG. Flexor tendon repair rehabilitation protocols: a systematic review. J Hand Surg Am. 2013;38(9):1712-7.e14.
- [Background] Caron Y. The real role of thumb in the overall function of hand. Sci Insights. 2025;47(3):1963-6.